CLINICAL TRIAL: NCT00336375
Title: Treatment of Uncomplicated Childhood Malaria by an Artemisinin Derivative in Combination With Lumefantrine. Efficacy, Safety and Genotyping.
Brief Title: Treatment of Uncomplicated Childhood Malaria in Tanzania by Artemether+Lumefantrine - Efficacy and Genotyping
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04/04/2006
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

ARMS (2):
- 1 (Experimental): All treatment doses accompanied with intake of fatty food
  Interventions: Drug: artemether-lumefantrine
- 2 (Active Comparator): All treatment doses not-accompanied with intake of fatty food.
  Interventions: Drug: artemether-lumefantrine

INTERVENTIONS:
Drug: artemether-lumefantrine — All treatment doses given either accompanied or not-accompanied with intake of fatty food.
  Other Names: All drug doses of artemether-lumefantrine is given either accompanied with or not-accompanied with intake of fatty food

SUMMARY:
The purpose of this explorative clinical trial is to study parasite population dynamics, diversity and clearance kinetics of Plasmodium falciparum as well as determination of the molecular mechanisms associated with drug resistance during the early phase of artemether-lumefantrine treatment when the drug intake is either accompanied with or without intake of fatty food. The hypothesis is that intake of fatty food together with artemether-lumefantrine will enhance parasite clearance and thereby decrease the risk of early selection of genetic markers related to drug resistance. The study population is children aged 1-10 years with uncomplicated malaria in Bagamoyo District, Tanzania. Enrolled children will be randomly allocated to either intake of a fatty meal or not together with the study drug. Artemether-lumefantrine will be given twice daily for 3 days in standard doses according to bodyweight. Study participants will be admitted during the study period (3 days)to allow close supervision and detailed blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-10 years
* Presence of asexual P. falciparum parasitaemia of 2000-200 000/μL
* No general danger signs or severe malaria present
* Haemoglobin ≥70 g/L
* History of fever within 24 hours OR axillary temperature ≥ 37.5Cº
* No other cause of fever is detectable
* No severe malnutrition
* Guardian/patient has understood the procedures of the study and willing to participate

Exclusion Criteria:

* Not able to drink or breastfeed
* Vomiting everything
* Recent history of convulsions
* Lethargic or unconscious
* Unable to sit or stand (as appropriate for age)
* History of allergy to test drugs
* History of intake of any drugs other than paracetamol and aspirin within 3 days
* Symptoms/signs of severe malaria

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2006-06; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Number of P.falciparum genotypes identified at baseline compared with accumulated number of genotypes in all blood samples | 72 hours

SECONDARY OUTCOMES:
Clearance kinetics of P. falciparum measured with PCR genotyping compared with blood slide reading | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anders Bjorkman, Professor, Study Director — Karolinska University Hospital
Locations (1):
- Fukayosi Primary Health Care Center, Fukayosi, Bagamoyo District, Tanzania

REFERENCES:
- [Derived] Mwaiswelo R, Ngasala B, Jovel I, Xu W, Larsson E, Malmberg M, Gil JP, Premji Z, Mmbando BP, Martensson A. Prevalence of and Risk Factors Associated with Polymerase Chain Reaction-Determined Plasmodium falciparum Positivity on Day 3 after Initiation of Artemether-Lumefantrine Treatment for Uncomplicated Malaria in Bagamoyo District, Tanzania. Am J Trop Med Hyg. 2019 May;100(5):1179-1186. doi: 10.4269/ajtmh.18-0729. PMID 30860013
- [Derived] Carlsson AM, Ngasala BE, Dahlstrom S, Membi C, Veiga IM, Rombo L, Abdulla S, Premji Z, Gil JP, Bjorkman A, Martensson A. Plasmodium falciparum population dynamics during the early phase of anti-malarial drug treatment in Tanzanian children with acute uncomplicated malaria. Malar J. 2011 Dec 20;10:380. doi: 10.1186/1475-2875-10-380. PMID 22185672